CLINICAL TRIAL: NCT01916252
Title: A Randomized, National, Open-label, Multicenter, Phase III Trial Studying Induction Therapy With Bortezomib/Lenalidomide/Dexamethasone (VRD-GEM), Followed by High-dose Chemotherapy With Melphalan-200 (MEL-200) Versus Busulfan-melphalan (BUMEL), and Consolidation With VRD-GEM in Patients Under 65 Years Old With Newly-diagnosed, Symptomatic Multiple Myeloma
Brief Title: Bortezomib (Velcade®), Lenalidomide (Revlimid®) and IV Busulfan (Busilvex®) in Patients Under 65 Years Old
Acronym: GEM2012MENOS65
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Collaborators: Janssen, LP (Industry); Celgene (Industry); Pierre Fabre Medicament (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEM2012MENOS65
Record Dates: First submitted 2013-07-30; First posted 2013-08-05 (Estimated); Last update posted 2017-09-27 (Actual); Status verified 2016-12

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; MEL200; BUMEL
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Lenalidomide; Busulfan; dexamethasone acetate; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MEL-200 (Active Comparator): bortezomib/lenalidomide/dexamethasone (VRD-GEM) induction treatment followed by high-dose melphalan-200 (MEL-200)
  Interventions: Drug: bortezomib (Velcade ®); Drug: lenalidomide (Revlimid®); Drug: Dexamethasone acetate; Drug: Melphalan
- BUMEL (Active Comparator): bortezomib/lenalidomide/dexamethasone (VRD-GEM) induction treatment followed by busulfan-melphalan (BUMEL) chemotherapy and consolidation with VRD-GEM
  Interventions: Drug: bortezomib (Velcade ®); Drug: lenalidomide (Revlimid®); Drug: busulfan (Busilvex ®); Drug: Dexamethasone acetate; Drug: Melphalan

INTERVENTIONS:
Drug: bortezomib (Velcade ®)
Drug: lenalidomide (Revlimid®)
Drug: busulfan (Busilvex ®)
  Arms: BUMEL
Drug: Dexamethasone acetate
Drug: Melphalan

SUMMARY:
This protocol is a national, multicenter, comparative, open-label, randomized trial comparing the progression free survival (PFS) of two pre-transplant conditioning regimens (BUMEL versus. MEL-200).

A total of 460 patients will be enrolled in the study. Scheduled evaluations and study visits will take place during the pre-treatment, treatment and follow-up periods.

The pre-treatment period includes the screening visit in which participants provide informed consent in writing in order to take part in the study. The patient is then assessed to determine his/her eligibility. The selection process will begin 21 days before the first dose of medication is administered (days -21 to 0). During the treatment period, eligible patients will be included in the study and given six cycles of induction treatment with bortezomib/ lenalidomide / dexamethasone (VRD-GEM). Each cycle will last 28 days, during which SC bortezomib will be administered on days 1, 4, 8 and 11, oral lenalidomide on days 1-21 of each cycle, and oral dexamethasone on days 1-4 and 9-12 of the cycle.

After the first three induction cycles, and in the absence of progression or unacceptable toxicity, peripheral blood hematopoietic stem cells will be mobilized and collected using G-CSF for later autologous transplantation. Patients will be randomized in a 1:1 allocation ratio to receive conditioning treatment with MEL-200 versus BUMEL. Randomization will take place at the beginning of the study, once the screening is complete and the patient's eligibility verified. Three months after transplantation, patients will receive two cycles of consolidation treatment with VRD-GEM at the same doses administered during induction treatment.

Once the treatment phase is complete, patients will begin the follow-up phase in which they will be visited every three months to evaluate disease progression and survival

ELIGIBILITY:
Inclusion Criteria:

* The patient must, in the opinion of the investigator, be capable of complying with all requirements of the trial
* Have signed the informed consent form
* Be between 18 and 65 years of age and a candidate for autologous stem cell transplant
* Have an ECOG Performance Status > 2 (or 3 if the ECOG is due to myeloma)
* Newly diagnosed patient with symptomatic multiple myeloma based on standard criteria, who has not received any prior chemotherapy treatment for Multiple Myeloma.
* Patient must have measurable disease, defined by the following criteria:

For secretory MM, measurable disease is defined by any quantifiable value of serum M-protein (IgG ≥ 10 g/L or IgA > 5 g/L) and/or, when applicable, an excretion of light chain in urine ≥ 200 mg/24 hours.

For oglio- or non-secretory multiple myeloma, measurable disease is defined by the presence of soft tissue (not bone) plasmacytomas, which is determined by clinical exam or radiographic techniques.

* Life expectancy > 3 months.
* The patient must have the following laboratory values in the 21 days prior to initiation of treatment (day 1, cycle 1):

Platelet count ≥ 100 x 109/L and absolute neutrophil count of ≥ 1.0 x 109/L Corrected serum calcium < 14 mg/dL. Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x the upper limit of normal (ULN).

Total bilirubin within normal limits. Serum creatinine ≤ 2 mg/dL

- Women of childbearing potential and men (including vasectomized men whose partners are women of childbearing potential), must use two methods of contraception during the entire course of treatment, during dose interruptions and for up to three months after receiving the final dose

Exclusion Criteria:

* Non-secretory myeloma without measurable plasmacytomas.
* Patients who have undergone prior treatment for multiple myeloma, with the exception of emergency treatment using steroid pulses, bisphosphonates, or radiotherapy received before beginning induction treatment.
* Peripheral neuropathy ≥ grade 2 in the 21 days prior to inclusion.
* Known hypersensitivity to bortezomib, boric acid, mannitol or lenalidomide.
* Patients that have received any investigational agent in the 28 days prior to inclusion in the study.
* Patients who have had a myocardial infarction in the six months prior to inclusion in this study or who are a class III or IV according to the New York Heart Association (NYHA) functional classification system, heart failure, unstable angina, uncontrolled ventricular arrhythmias or acute ischemia detected by electrocardiogram, or nervous system disorders.
* Patients currently enrolled in another clinical trial or receiving any type of investigational agent.
* Patients who are seropositive for HBV, HCV or HIV.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2013-09; Primary Completion 2016-11-16 (Actual); Study Completion 2016-11-16 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival to measure the treatment efficacy | 2 years

SECONDARY OUTCOMES:
Complete response rates to measure the treatment efficacy | 1 year
Evaluation of minimal residual disease immunofixation negative-CR after each phase of treatment | 1 year
Overall survival | Time to death
Describe the adverse events to evaluate the safety and tolerability | 4 years

CONTACTS AND LOCATIONS:
Locations (74):
- Spain (74):
  - Hospital Son Espases (Son Dureta), Mallorca, Balearic Islands
  - Hospital Son Llátzer, Palma de Mallorca, Balearic Islands
  - Hospital Durán i Reynals - ICO L´Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - H. Althaia, Xarxa Asistencial de Manresa, Manresa, Barcelona
  - Hospital de Gran Canaria Dr. Negrín, Las Palmas de Gran Canaria, Canary Islands
  - Hospital Esp. de Jerez de la Frontera, Jerez de la Frontera, Cádiz
  - Hospital Nuestra Señora del Prado, Talavera de La Reina, Madrid
  - Complejo Universitario de Toledo, Toledo, Madrid
  - Hospital General de Albacete, Albacete
  - Hospital Univ. Fundación de Alcorcón, Alcorcón
  - Hospital General Univ. de Alicante, Alicante
  - Hospital Torrevieja Salud UTE, Alicante
  - Hospital del Tajo, Aranjuez
  - Hospital German Trias i Pujol, Badalona
  - Hospital de Cruces, Barakaldo
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Vall d´Hebrón, Barcelona
  - Hospital Universitario de Burgos, Burgos
  - Hospital General Univ. Santa Lucía, Cartagena
  - Hospital General de Castellón, Castellon
  - Hospital San Pedro de Alcántara (Complejo Hospitalario de Cáceres), Cáceres
  - Hospital General de Ciudad Real, Ciudad Real
  - Hospital del Vinalopó, Elche
  - Hospital de Fuenlabrada, Fuenlabrada
  - Hospital de Cabueñes, Gijón
  - H. Univ. de Girona Dr. Josep Trueta (ICO), Girona
  - Complejo Hosp. Virgen de las Nieves, Granada
  - Hospital Universitario de Guadalajara, Guadalajara
  - Hospital Severo Ochoa, Leganés
  - Hospital de León, León
  - Hospital Universitari Arnau de Vilanova de Lleida, Lleida
  - Hospital San Pedro, Logroño
  - Centro Oncológico MD Anderson, Madrid
  - Fundación Jiménez Díaz-UTE, Madrid
  - Hospital Clínico Universitario San Carlos, Madrid
  - Hospital General Univ. Gregorio Marañón, Madrid
  - Hospital Infanta Cristina, Madrid
  - Hospital Infanta Leonor, Madrid
  - Hospital Infanta Sofía, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Madrid Sanchinarro, Madrid
  - Hospital Universitario Puerta de Hierro-Majadahonda, Majadahonda
  - Complejo Hospitalario Costa del Sol, Marbella
  - Hospital Morales Meseguer, Murcia
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Complejo Hospitalario Ourense, Ourense
  - Hospital Universitario Central Asturias, Oviedo
  - Clínica Universidad de Navarra, Pamplona
  - Complejo Hospitalario de Navarra (Hospital Virgen del Camino), Pamplona
  - Complejo Hospitalario Pontevedra, Pontevedra
  - Hospital de Sabadell (Parc Taulí), Sabadell
  - Hospital Clínico de Salamanca, Salamanca
  - Hospital Universitario de Donostia, San Sebastián
  - Hospital Univ. Marqués de, Santander
  - Complejo Universitario de Santiago, Santiago de Compostela
  - Hospital General de Segovia, Segovia
  - Complejo Hosp. Regional Virgen del Rocío, Seville
  - Hospital Nuestra Señora de Valme, Seville
  - Hospital Santa Bárbara, Soria
  - H. Universitari de Tarragona Joan XXIII, Tarragona
  - Hospital Universitari Mutua de Terrassa, Terrassa
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario Dr. Peset, Valencia
  - Hospital Universitario La Fe, Valencia
  - Hospital Clínico de Valladolid, Valladolid
  - Hospital Universitario Río Hortega, Valladolid
  - Hospital de Txagorritxu, Vitoria-Gasteiz
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza
  - Hospital Miguel Servet, Zaragoza

REFERENCES:
- [Derived] Lahuerta JJ, San-Miguel J, Jimenez-Ubieto A, Alonso R, Paiva B, Puig N, Cedena MT, Gutierrez NC, Calasanz MJ, Fernandez Guijarro M, Tamayo RR, Rocafiguera AO, Blanchard MJ, Carrillo Cruz E, Martinez-Martinez R, Bargay J, Sureda Balari A, Rubia J, Hernandez Garcia MT, Cabanas V, Montero FC, Bernal LP, Montes YG, Martinez-Lopez J, Rodriguez-Otero P, Krisnik I, Arguinano JM, Gonzalez Garcia ME, Ocio EM, Cruz J, Mateos MV, Rosinol L, Blade J. High-dose busulfan-melphalan vs melphalan and reinforced VRD for newly diagnosed multiple myeloma: a phase 3 GEM trial. Blood. 2025 Oct 9;146(15):1747-1758. doi: 10.1182/blood.2025028313. PMID 40499010
- [Derived] Puig N, Agullo C, Contreras T, Cedena MT, Martinez-Lopez J, Oriol A, Blanchard MJ, Rios R, Inigo MB, Sureda A, Lakhwani S, de la Rubia J, Gonzalez-Calle V, Cabanas V, Palomera L, Moraleda JM, Bargay J, Castro S, Rosinol L, Blade J, San-Miguel JF, Lahuerta JJ, Paiva B, Mateos MV. Measurable residual disease by mass spectrometry and next-generation flow to assess treatment response in myeloma. Blood. 2024 Dec 5;144(23):2432-2438. doi: 10.1182/blood.2024024995. PMID 39293025
- [Derived] Guerrero C, Puig N, Cedena MT, Calasanz MJ, Gutierrez NC, Fernandez M, Oriol A, Rios-Tamayo R, Hernandez MT, Martinez-Martinez R, Bargay J, de Arriba F, Palomera L, Gonzalez-Rodriguez AP, Gonzalez Perez MS, Orfao A, Mateos MV, Martinez-Lopez J, Rosinol L, Blade J, Lahuerta JJ, San-Miguel JF, Paiva B. Predictors of unsustained measurable residual disease negativity in transplant-eligible patients with multiple myeloma. Blood. 2024 Feb 15;143(7):597-603. doi: 10.1182/blood.2023022083. PMID 38048552
- [Derived] Lakhwani S, Rosinol L, Puig N, Pico-Picos MA, Medina-Gonzalez L, Martinez-Lopez J, Paiva B, Cedena MT, Oriol A, Rios-Tamayo R, Blanchard MJ, Jarque I, Bargay J, Moraleda JM, Carrillo-Cruz E, Sureda A, Krsnik I, Gonzalez E, Casado LF, Marti JM, Encinas C, De Arriba F, Palomera L, Sampol A, Gonzalez-Montes Y, Motllo C, De La Cruz J, Alonso R, Mateos MV, Blade J, Lahuerta JJ, San-Miguel J, Hernandez MT. Recovery of uninvolved heavy/light chain pair immunoparesis in newly diagnosed transplant-eligible myeloma patients complements the prognostic value of minimal residual disease detection. Haematologica. 2024 Jun 1;109(6):1909-1917. doi: 10.3324/haematol.2023.284154. PMID 38031761
- [Derived] Rosinol L, Hebraud B, Oriol A, Colin AL, Rios Tamayo R, Hulin C, Blanchard MJ, Caillot D, Sureda A, Hernandez MT, Arnulf B, Mateos MV, Macro M, San-Miguel J, Belhadj K, Lahuerta JJ, Garelik MB, Blade J, Moreau P. Integrated analysis of randomized controlled trials evaluating bortezomib + lenalidomide + dexamethasone or bortezomib + thalidomide + dexamethasone induction in transplant-eligible newly diagnosed multiple myeloma. Front Oncol. 2023 Nov 2;13:1197340. doi: 10.3389/fonc.2023.1197340. eCollection 2023. PMID 38023148
- [Derived] Cardona-Benavides IJ, Misiewicz-Krzeminska I, Rojas EA, De Ramon C, Sanz-Solas A, Isidro I, Quwaider D, Lopez-Guerrero AM, Cuadrado M, Calasanz MJ, Rosinol L, Martinez-Lopez J, San Miguel JF, Mateos MV, Corchete LA, Gutierrez NC. Quantification of cyclin D1 and D2 proteins in multiple myeloma identifies different expression patterns from those revealed by gene expression profiling. Haematologica. 2024 Mar 1;109(3):877-887. doi: 10.3324/haematol.2023.283445. PMID 37646661
- [Derived] Puig N, Contreras MT, Agullo C, Martinez-Lopez J, Oriol A, Blanchard MJ, Rios R, Martin J, Inigo MB, Sureda A, Hernandez MT, de la Rubia J, Gonzalez-Calle V, Krsnik I, Cabanas V, Palomera L, Moraleda JM, Bargay J, Cedena MT, Paiva B, Rosinol L, Blade J, San Miguel J, Lahuerta JJ, Mateos MV. Mass spectrometry vs immunofixation for treatment monitoring in multiple myeloma. Blood Adv. 2022 Jun 14;6(11):3234-3239. doi: 10.1182/bloodadvances.2021006762. PMID 35157768
- [Derived] Botta C, Maia C, Garces JJ, Termini R, Perez C, Manrique I, Burgos L, Zabaleta A, Alignani D, Sarvide S, Merino J, Puig N, Cedena MT, Rossi M, Tassone P, Gentile M, Correale P, Borrello I, Terpos E, Jelinek T, Paiva A, Roccaro A, Goldschmidt H, Avet-Loiseau H, Rosinol L, Mateos MV, Martinez-Lopez J, Lahuerta JJ, Blade J, San-Miguel JF, Paiva B. FlowCT for the analysis of large immunophenotypic data sets and biomarker discovery in cancer immunology. Blood Adv. 2022 Jan 25;6(2):690-703. doi: 10.1182/bloodadvances.2021005198. PMID 34587246
- [Derived] Goicoechea I, Puig N, Cedena MT, Burgos L, Cordon L, Vidriales MB, Flores-Montero J, Gutierrez NC, Calasanz MJ, Ramos MM, Lara-Astiaso D, Vilas-Zornoza A, Alignani D, Rodriguez I, Sarvide S, Alameda D, Garces JJ, Rodriguez S, Fresquet V, Celay J, Garcia-Sanz R, Martinez-Lopez J, Oriol A, Rios R, Martin-Sanchez J, Martinez-Martinez R, Sarra J, Hernandez MT, de la Rubia J, Krsnik I, Moraleda JM, Palomera L, Bargay J, Martinez-Climent JA, Orfao A, Rosinol L, Mateos MV, Lahuerta JJ, Blade J, San Miguel J, Paiva B. Deep MRD profiling defines outcome and unveils different modes of treatment resistance in standard- and high-risk myeloma. Blood. 2021 Jan 7;137(1):49-60. doi: 10.1182/blood.2020006731. PMID 32693406
- [Derived] Rosinol L, Oriol A, Rios R, Sureda A, Blanchard MJ, Hernandez MT, Martinez-Martinez R, Moraleda JM, Jarque I, Bargay J, Gironella M, de Arriba F, Palomera L, Gonzalez-Montes Y, Marti JM, Krsnik I, Arguinano JM, Gonzalez ME, Gonzalez AP, Casado LF, Lopez-Anglada L, Paiva B, Mateos MV, San Miguel JF, Lahuerta JJ, Blade J. Bortezomib, lenalidomide, and dexamethasone as induction therapy prior to autologous transplant in multiple myeloma. Blood. 2019 Oct 17;134(16):1337-1345. doi: 10.1182/blood.2019000241. PMID 31484647